CLINICAL TRIAL: NCT03833661
Title: A Phase II, Multicenter, Open-label Study to Investigate the Clinical Efficacy of M7824 Monotherapy in Participants With Locally Advanced or Metastatic Biliary Tract Cancer Who Fail or Are Intolerant to First-line Platinum-Based Chemotherapy
Brief Title: M7824 Monotherapy in Locally Advanced or Metastatic Second Line (2L) Biliary Tract Cancer (Cholangiocarcinoma and Gallbladder Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200647_0047; 2018-003707-19 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer
Keywords: M7824; Bintrafusp alfa (proposed INN); Transforming growth factor-beta; First-line Platinum-Based Chemotherapy; Programmed death-ligand 1; Metastatic Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms; Camurati-Engelmann Syndrome | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M7824 (Experimental)
  Interventions: Drug: M7824

INTERVENTIONS:
Drug: M7824 — Participants received an intravenous infusion of 1200 milligrams (mg) M7824 once every 2 weeks until confirmed disease progression, death, unacceptable toxicity or study withdrawal.
  Other Names: Bintrafusp alfa

SUMMARY:
The study to evaluate M7824 monotherapy in participants with advanced or metastatic biliary tract cancer (BTC) who failed or were intolerant to first-line (1L) chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Are participants with histologically or cytologically confirmed locally advanced or metastatic BTC.
* Availability of tumor (primary or metastatic) archival material or fresh biopsies is mandatory
* Participants with BTC must have failed or be intolerant to 1L systemic platinum-based chemotherapy administered for locally advanced or metastatic disease. Only one prior treatment line is allowed
* Disease must be measurable with at least 1 unidimensionally measurable lesion by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 1
* Life expectancy >= 12 weeks as judged by the Investigator
* Adequate hematological function defined by white blood cell (WBC) count >= 3 * 10^9/Litre with absolute neutrophil count (ANC) >= 1.5 * 109/Litre, lymphocyte count >= 0.5 * 10^9/Litre, platelet count >=75 * 10^9/Litre, and hemoglobin (Hgb) >= 9 grams/decilitre
* Adequate hepatic function defined by a total bilirubin level =< 1.5 * upper limit of normal (ULN), an aspartate aminotransferase (AST) level =< 2.5 * ULN, and an alanine aminotransferase (ALT) level =<2.5 * ULN. For participants with liver involvement in their tumor, AST =< 5.0 * ULN and ALT =< 5.0 * ULN is acceptable
* Adequate coagulation function defined as prothrombin time (PT) or international normalized ratio (INR) =< 1.5 * ULN unless the participant is receiving anticoagulant therapy
* Albumin >= 3.0 grams/decilitre
* Hepatitis B virus (HBV) deoxyribonucleic acid (DNA) positive participants must be treated and on a stable dose of antivirals
* Adequate renal function defined by either creatinine =< 1.5 * ULN or an estimated creatinine clearance (CCr) > 40 milliliter (mL) per minute (min) according to the Cockcroft-Gault formula or by measure of CCr from 24-hour urine collection
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Ampullary cancer was excluded
* Significant acute or chronic infections
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Interstitial lung disease or its history
* Participants who were not eligible for or have not been treated with 1L systemic chemotherapy
* Anticancer treatment within 21 days before the start of study intervention
* Concurrent treatment with nonpermitted drugs
* Prior participation in a M7824 clinical trial
* Prior therapy with other immunotherapy or checkpoint inhibitors, such as anti-PD 1, anti PD L1, anti- cytotoxic T-cell lymphocyte-4 (CTLA-4) antibodies.
* Pregnancy or breast feeding
* Systemic anticancer treatment after failing 1L platinum-based chemotherapy
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (33):
- United States (7):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - UCSF Mount Zion Medical Ctr, San Francisco, California
  - Mayo Clinic in Florida - Department of Neurology, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - MD Anderson Cancer Center - Unit, Houston, Texas
- China (2):
  - Peking University Cancer Hospital, Beijing
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin
- France (3):
  - Groupe Hospitalier Sud - Hôpital Haut Lévêque - Service Hepato Gastroentérologie Oncologie Digest, Pessac
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Italy (4):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi - Unita' Operativa di Pediatria, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori Milano, Milan
  - Policlinico Universitario Agostino Gemelli - UOC Oncologia Medica, Roma
- Japan (5):
  - National Cancer Center Hospital - Dept of Hepatobiliary and Pancreatic Oncology, Chūōku
  - National Cancer Center Hospital East, Kashiwa-shi
  - Kyorin University Hospital - Dept of Oncology, Mitaka-shi
  - Kindai University Hospital - Dept of Gastroenterology, Osakasayama-shi
  - Kanagawa Cancer Center, Yokohama
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
- Taiwan (3):
  - Chang Gung Memorial Hospital, Linkou, Linkou District
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- St James's University Hospital - Dept of Oncology, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Yoo C, Oh DY, Choi HJ, Kudo M, Ueno M, Kondo S, Chen LT, Osada M, Helwig C, Dussault I, Ikeda M. Phase I study of bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1, in patients with pretreated biliary tract cancer. J Immunother Cancer. 2020 May;8(1):e000564. doi: 10.1136/jitc-2020-000564. PMID 32461347
- [Derived] Milenkovic-Grisic AM, Terranova N, Mould DR, Vugmeyster Y, Mrowiec T, Machl A, Girard P, Venkatakrishnan K, Khandelwal A. Tumor growth inhibition modeling in patients with second line biliary tract cancer and first line non-small cell lung cancer based on bintrafusp alfa trials. CPT Pharmacometrics Syst Pharmacol. 2024 Jan;13(1):143-153. doi: 10.1002/psp4.13068. Epub 2023 Dec 13. PMID 38087967
- [Derived] Yoo C, Javle MM, Verdaguer Mata H, de Braud F, Trojan J, Raoul JL, Kim JW, Ueno M, Lee CK, Hijioka S, Cubillo A, Furuse J, Azad N, Sato M, Vugmeyster Y, Machl A, Bajars M, Bridgewater J, Oh DY, Borad MJ. Phase 2 trial of bintrafusp alfa as second-line therapy for patients with locally advanced/metastatic biliary tract cancers. Hepatology. 2023 Sep 1;78(3):758-770. doi: 10.1097/HEP.0000000000000365. Epub 2023 Apr 1. PMID 36999533
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200647_0047
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First participant signed informed consent: 26 Mar 2019, Clinical cutoff date: 30 March 2021.
Groups:
- M7824: Participants received intravenous infusion of M7824 at a dose of 1200 milligrams (mg) once every 2 weeks until confirmed progression of disease, death, unacceptable toxicity, or study withdrawal.
Period: Overall Study
Arm/Group | M7824
Started | 159
Completed | 159
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) analysis set included all participants who were administered at least one dose of M7824.
Arm/Group | M7824
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 155
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 77
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 64
  More than one race | 0
  Unknown or Not Reported | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: Confirmed objective response was defined as the percentage of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by IRC.
Time Frame: Time from first treatment up to 555 days
Population: ITT analysis set included all participants who were administered at least one dose of M7824.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 159
percentage of participants | 10.7 [6.4 to 16.6]

2. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by IRC. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Time from first documentation of objective response to data cutoff (assessed up to 736 days)
Population: ITT analysis set included all participants who were administered at least one dose of M7824. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 17
months | 10.0 [3.9 to NA] — The upper limit could not be estimated due to insufficient number of events by the date of data cutoff.

3. Secondary Outcome: Durable Response Rate (DRR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC)
Description: DRR was defined as the percentage of participants with confirmed objective response (CR or PR) with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DRR was determined according to RECIST v1.1 and assessed by IRC.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 17
percentage of participants | 6.3 [3.1 to 11.3]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs, Including Adverse Event of Special Interests (AESIs)
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious AEs and non-serious AEs. Treatment-related TEAEs: reasonably related to the study intervention. AESIs included Infusion-related reactions, Immune-related AEs, Transforming growth factor-beta (TGF-β) inhibition mediated skin AE and anemia.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: Safety analysis set included all participants who were administered at least one dose of M7824.
Measure: Count of Participants; unit: Participants
Arm/Group | M7824
Number analyzed (Participants) | 159
Participants
  TEAEs | 152
  Treatment Related TEAEs | 99
  AESI: Infusion-related reaction | 10
  AESI: Immune-related AE | 46
  AESI: TGF-β inhibition mediated skin AE | 13
  AESI: Anemia | 44

5. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) Assessed by Independent Review Committee (IRC)
Description: PFS was defined as the time from first administration of study intervention until the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first administration of study drug until the first documentation of PD or death, assessed up to data-cutoff (736 days)
Population: ITT analysis set included all participants who were administered at least one dose of M7824.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 159
months | 1.8 [1.7 to 1.8]

6. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: Confirmed objective response was defined as the percentage of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by Investigator.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: ITT analysis set included all participants who were administered at least one dose of M7824.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 159
percentage of participants | 10.7 [6.4 to 16.6]

7. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Rresponse [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) and assessed by Investigator. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Time from first documentation of objective response to data cutoff (assessed up to 736 days)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 17
months | 8.2 [3.9 to 12.0]

8. Secondary Outcome: Durable Response Rate (DRR) Acoording to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: DRR was defined as the percentage of participants with confirmed objective response (CR or PR) with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DRR was determined according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) and assessed by Investigator.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 17
percentage of participants | 5.7 [2.6 to 10.5]

9. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by the Investigator
Description: as for outcome 5
Time Frame: as for outcome 5
Population: ITT analysis set included all participants who were administered at least one dose of M7824.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 159
months | 1.8 [1.7 to 1.8]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from first administration of study intervention to the date of death due to any cause. The OS was analyzed by using the Kaplan-Meier method.
Time Frame: Time from first administration of study drug to data cutoff (assessed up to 736 days)
Population: ITT analysis set included all participants who were administered at least one dose of M7824.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 159
months | 7.6 [5.8 to 9.5]

11. Secondary Outcome: Serum Pre-Dose Concentrations (Ctrough) of M7824
Description: Ctrough was defined as the concentration observed immediately before next dosing (corresponding to pre-dose or trough concentration for multiple dosing).
Time Frame: At Day 15, Day 29, Day 43, Day 85, Day 127, Day 169, Day 253, Day 337, Day 421 and Day 505
Population: Pharmacokinetic (PK) analysis set included all participants who completed at least one dose of M7824 and who provided at least one sample with a measurable concentration of M7824. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | M7824
Number analyzed (Participants) | 138
microgram per milliliter (mcg/mL)
  Day 15 | 70.7 (40.7)
  Day 29: number analyzed (Participants) | 105
  Day 29 | 84.2 (58.0)
  Day 43: number analyzed (Participants) | 89
  Day 43 | 93.4 (52.6)
  Day 85: number analyzed (Participants) | 40
  Day 85 | 105 (42.6)
  Day 127: number analyzed (Participants) | 26
  Day 127 | 117 (41.5)
  Day 169: number analyzed (Participants) | 12
  Day 169 | 101 (55.6)
  Day 253: number analyzed (Participants) | 13
  Day 253 | 115 (46.8)
  Day 337: number analyzed (Participants) | 6
  Day 337 | 91.3 (41.5)
  Day 421: number analyzed (Participants) | 5
  Day 421 | 114 (36.7)
  Day 505: number analyzed (Participants) | 2
  Day 505 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated if fewer than 3 participants have reportable parameter values.

12. Secondary Outcome: Serum Concentration at End of Infusion (CEOI) of M7824
Description: Serum Concentration at End of Infusion (CEOI) of M7824 is reported.
Time Frame: At Day 1 and Day 29
Population: PK analysis set included all participants who completed at least one dose of M7824 and who provided at least one sample with a measurable concentration of M7824. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | M7824
Number analyzed (Participants) | 152
mcg/mL
  Day 1 | 399 (31.5)
  Day 29: number analyzed (Participants) | 104
  Day 29 | 434 (48.5)

13. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA)
Description: Serum samples were analyzed by a validated assay method to detect the presence of antidrug antibodies (ADA). Number of participants with positive ADA were reported.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: Immunogenicity analysis set included all participants who received at least one dose of M7824 and who had at least one valid result of ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | M7824
Number analyzed (Participants) | 157
Participants | 45

14. Secondary Outcome: Percentage of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Independent Review Committee (IRC) According to Programmed Death Ligand 1 (PD-L1) Expression
Description: Confirmed objective response was defined as the percentage of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed objective response was determined according to RECIST v1.1 and as adjudicated by IRC through PD-L1 Subgroup: PD-L1 expression on tumor cells (TC) and on immune cells (IC) at baseline and in the following categories: <1%, >=1%, <5%, >=5%, <25%, >=25%, <50%, >=50% were reported.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: ITT analysis set included all participants who were administered at least one dose of M7824. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable for the specified categories for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 141
percentage of participants
  PD-L1 expression on TC: < 1%: number analyzed (Participants) | 98
  PD-L1 expression on TC: < 1% | 10.2 [5.0 to 18.0]
  PD-L1 expression on TC: >= 1%: number analyzed (Participants) | 43
  PD-L1 expression on TC: >= 1% | 7.0 [1.5 to 19.1]
  PD-L1 expression on TC: < 5%: number analyzed (Participants) | 113
  PD-L1 expression on TC: < 5% | 9.7 [5.0 to 16.8]
  PD-L1 expression on TC: >= 5%: number analyzed (Participants) | 28
  PD-L1 expression on TC: >= 5% | 7.1 [0.9 to 23.5]
  PD-L1 expression on TC: < 25%: number analyzed (Participants) | 126
  PD-L1 expression on TC: < 25% | 8.7 [4.4 to 15.1]
  PD-L1 expression on TC: >= 25%: number analyzed (Participants) | 15
  PD-L1 expression on TC: >= 25% | 13.3 [1.7 to 40.5]
  PD-L1 expression on TC: < 50%: number analyzed (Participants) | 130
  PD-L1 expression on TC: < 50% | 9.2 [4.9 to 15.6]
  PD-L1 expression on TC: >= 50%: number analyzed (Participants) | 11
  PD-L1 expression on TC: >= 50% | 9.1 [0.2 to 41.3]
  PD-L1 expression on IC: < 1%: number analyzed (Participants) | 22
  PD-L1 expression on IC: < 1% | 13.6 [2.9 to 34.9]
  PD-L1 expression on IC: >= 1%: number analyzed (Participants) | 108
  PD-L1 expression on IC: >= 1% | 7.4 [3.3 to 14.1]
  PD-L1 expression on IC: < 5%: number analyzed (Participants) | 46
  PD-L1 expression on IC: < 5% | 8.7 [2.4 to 20.8]
  PD-L1 expression on IC: >= 5%: number analyzed (Participants) | 84
  PD-L1 expression on IC: >= 5% | 8.3 [3.4 to 16.4]
  PD-L1 expression on IC: < 25%: number analyzed (Participants) | 120
  PD-L1 expression on IC: < 25% | 7.5 [3.5 to 13.8]
  PD-L1 expression on IC: >= 25%: number analyzed (Participants) | 10
  PD-L1 expression on IC: >= 25% | 20.0 [2.5 to 55.6]
  PD-L1 expression on IC: < 50%: number analyzed (Participants) | 129
  PD-L1 expression on IC: < 50% | 8.5 [4.3 to 14.7]
  PD-L1 expression on IC: >= 50%: number analyzed (Participants) | 1
  PD-L1 expression on IC: >= 50% | 0.0 [0.0 to 97.5]

15. Secondary Outcome: Percentage of Participants With Confirmed Objective Response as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Independent Review Committee (IRC) According to Microsatellite Instability (MSI) Status
Description: Confirmed OR was defined as the percentage of participants with a confirmed OR of CR or PR. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR). Confirmed OR was determined according to RECIST v1.1 and as adjudicated by IRC through MSI Status subgroups as:- MSI High = if participant is MSI High for any (at least one) test;- Microsatellite stable (MSS) or MSI Low = if participant is not MSI High for any test;- Unknown (missing) = no MSI tests available at baseline was reported. MSI high: if 2 or more unstable markers were detected in sample; MSI low: if 1 marker was unstable and remaining markers were stable and MSS if all markers were stable.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 153
percentage of participants
  High: number analyzed (Participants) | 3
  High | 0.0 [0.0 to 70.8]
  Low or Microsatellite stable: number analyzed (Participants) | 150
  Low or Microsatellite stable | 10.0 [5.7 to 16.0]
  Unknown (missing): number analyzed (Participants) | 0

16. Secondary Outcome: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by an Independent Review Committee (IRC) According to Programmed Death Ligand 1 (PD-L1) Expression
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and as adjudicated by IRC through PD-L1 Subgroup: PD-L1 expression on tumor cells (TC) and on immune cells (IC) at baseline and in the following categories: <1%, >=1%, <5%, >=5%, <25%, >=25%, <50%, >=50% was reported.
Time Frame: Time from first documentation of objective response to data cutoff (assessed up to 736 days)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 13
months
  PD-L1 expression on TC: < 1%: number analyzed (Participants) | 10
  PD-L1 expression on TC: < 1% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: >= 1%: number analyzed (Participants) | 3
  PD-L1 expression on TC: >= 1% | 5.8 [3.9 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: < 5%: number analyzed (Participants) | 11
  PD-L1 expression on TC: < 5% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: >= 5%: number analyzed (Participants) | 2
  PD-L1 expression on TC: >= 5% | NA [3.9 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: < 25%: number analyzed (Participants) | 11
  PD-L1 expression on TC: < 25% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: >= 25%: number analyzed (Participants) | 2
  PD-L1 expression on TC: >= 25% | NA [3.9 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: < 50%: number analyzed (Participants) | 12
  PD-L1 expression on TC: < 50% | NA [3.7 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on TC: >= 50%: number analyzed (Participants) | 1
  PD-L1 expression on TC: >= 50% | NA [NA to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: < 1%: number analyzed (Participants) | 3
  PD-L1 expression on IC: < 1% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: >= 1%: number analyzed (Participants) | 8
  PD-L1 expression on IC: >= 1% | NA [3.7 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: < 5%: number analyzed (Participants) | 4
  PD-L1 expression on IC: < 5% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: >= 5%: number analyzed (Participants) | 7
  PD-L1 expression on IC: >= 5% | NA [3.9 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: < 25%: number analyzed (Participants) | 9
  PD-L1 expression on IC: < 25% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: >= 25%: number analyzed (Participants) | 2
  PD-L1 expression on IC: >= 25% | NA [NA to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: < 50%: number analyzed (Participants) | 11
  PD-L1 expression on IC: < 50% | NA [3.4 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  PD-L1 expression on IC: >= 50%: number analyzed (Participants) | 0

17. Secondary Outcome: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by an Independent Review Committee (IRC) According to According to Microsatellite Instability (MSI) Status
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (CR) or (PR) to the date of first documentation of PD or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and as adjudicated by IRC through MSI Status subgroups as:- MSI High = if participant is MSI High for any (at least one) test;- MSS or MSI Low = if participant is not MSI High for any test;- Unknown (missing) = no MSI tests available at baseline was reported. MSI high: if 2 or more unstable markers were detected in sample; MSI low: if 1 marker was unstable and remaining markers were stable and MSS if all markers were stable.
Time Frame: Time from first documentation of objective response to data cutoff (assessed up to 736 days)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | M7824
Number analyzed (Participants) | 15
months
  High: number analyzed (Participants) | 0
  Low or Microsatellite stable | NA [3.7 to NA] — Due to small number of events, Median and Upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not derive.
  Unknown (missing): number analyzed (Participants) | 0

18. Secondary Outcome: Durable Response Rate (DRR) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by an Independent Review Committee (IRC) According to Programmed Death Ligand 1 (PD-L1) Expression
Description: DRR was defined as the percentage of participants with confirmed objective response (CR or PR) with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DRR was determined according to RECIST v1.1 and adjudicated by IRC through PD-L1 Subgroup: PD-L1 expression on tumor cells (TC) and on immune cells (IC) at baseline and in the following categories: <1%, >=1%, <5%, >=5%, <25%, >=25%, <50%, >=50% was reported.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 141
percentage of participants
  PD-L1 expression on TC: < 1%: number analyzed (Participants) | 98
  PD-L1 expression on TC: < 1% | 6.1 [2.3 to 12.9]
  PD-L1 expression on TC: >= 1%: number analyzed (Participants) | 43
  PD-L1 expression on TC: >= 1% | 2.3 [0.1 to 12.3]
  PD-L1 expression on TC: < 5%: number analyzed (Participants) | 113
  PD-L1 expression on TC: < 5% | 5.3 [2.0 to 11.2]
  PD-L1 expression on TC: >= 5%: number analyzed (Participants) | 28
  PD-L1 expression on TC: >= 5% | 3.6 [0.1 to 18.3]
  PD-L1 expression on TC: < 25%: number analyzed (Participants) | 126
  PD-L1 expression on TC: < 25% | 4.8 [1.8 to 10.1]
  PD-L1 expression on TC at >= 25%: number analyzed (Participants) | 15
  PD-L1 expression on TC at >= 25% | 6.7 [0.2 to 31.9]
  PD-L1 expression on TC: < 50%: number analyzed (Participants) | 130
  PD-L1 expression on TC: < 50% | 4.6 [1.7 to 9.8]
  PD-L1 expression on TC: >= 50%: number analyzed (Participants) | 11
  PD-L1 expression on TC: >= 50% | 9.1 [0.2 to 41.3]
  PD-L1 expression on IC: < 1%: number analyzed (Participants) | 22
  PD-L1 expression on IC: < 1% | 9.1 [1.1 to 29.2]
  PD-L1 expression on IC: >= 1%: number analyzed (Participants) | 108
  PD-L1 expression on IC: >= 1% | 3.7 [1.0 to 9.2]
  PD-L1 expression on IC: < 5%: number analyzed (Participants) | 46
  PD-L1 expression on IC: < 5% | 4.3 [0.5 to 14.8]
  PD-L1 expression on IC: >= 5%: number analyzed (Participants) | 84
  PD-L1 expression on IC: >= 5% | 4.8 [1.3 to 11.7]
  PD-L1 expression on IC: < 25%: number analyzed (Participants) | 120
  PD-L1 expression on IC: < 25% | 3.3 [0.9 to 8.3]
  PD-L1 expression on IC: >= 25%: number analyzed (Participants) | 10
  PD-L1 expression on IC: >= 25% | 20.0 [2.5 to 55.6]
  PD-L1 expression on IC: < 50%: number analyzed (Participants) | 129
  PD-L1 expression on IC: < 50% | 4.7 [1.7 to 9.8]
  PD-L1 expression on IC: >= 50%: number analyzed (Participants) | 1
  PD-L1 expression on IC: >= 50% | 0.0 [0.0 to 97.5]

19. Secondary Outcome: Durable Response Rate (DRR) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by an Independent Review Committee (IRC) According to According to Microsatellite Instability (MSI) Status
Description: DRR was defined as the percentage of participants with confirmed OR (CR or PR) with duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DRR was determined according to RECIST v1.1 and adjudicated by IRC through MSI Status subgroups as:- MSI High = if participant is MSI High for any (at least one) test;- MSS or MSI Low = if participant is not MSI High for any test;- Unknown (missing) = no MSI tests available at baseline was reported. MSI high: if 2 or more unstable markers were detected in sample; MSI low: if 1 marker was unstable and remaining markers were stable and MSS if all markers were stable.
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | M7824
Number analyzed (Participants) | 153
percentage of participants
  High: number analyzed (Participants) | 3
  High | 0.0 [0.0 to 70.8]
  Low or Microsatellite stable: number analyzed (Participants) | 150
  Low or Microsatellite stable | 4.0 [1.5 to 8.5]
  Unknown (missing): number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Time from first treatment to data cutoff (assessed up to 736 days)
Arm/Group | M7824
All-Cause Mortality (participants affected / at risk) | 108/159
Serious Adverse Events (participants affected / at risk) | 86/159
Other Adverse Events (participants affected / at risk) | 144/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M7824 (N=159)
Anaemia (Blood and lymphatic system disorders) | 5
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Myocarditis (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Duodenal stenosis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric stenosis (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Disease progression (General disorders) | 16
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 3
Bile duct stenosis (Hepatobiliary disorders) | 3
Cholangitis (Hepatobiliary disorders) | 8
Cholangitis acute (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 4
Hepatitis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 3
Liver injury (Hepatobiliary disorders) | 2
Abdominal infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 6
Bursitis infective (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Infective spondylitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Staphylococcal infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Varicella zoster pneumonia (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Vascular device infection (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour hyperprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Immune-mediated encephalitis (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Nephritis (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Biliary stent placement (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M7824 (N=159)
Anaemia (Blood and lymphatic system disorders) | 41
Hypothyroidism (Endocrine disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 21
Ascites (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 23
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 23
Fatigue (General disorders) | 23
Oedema peripheral (General disorders) | 11
Pyrexia (General disorders) | 25
Infusion related reaction (Injury, poisoning and procedural complications) | 8
Alanine aminotransferase increased (Investigations) | 24
Aspartate aminotransferase increased (Investigations) | 26
Blood alkaline phosphatase increased (Investigations) | 17
Blood bilirubin increased (Investigations) | 16
Decreased appetite (Metabolism and nutrition disorders) | 34
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16
Hyponatraemia (Metabolism and nutrition disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 11
Headache (Nervous system disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 29
Rash (Skin and subcutaneous tissue disorders) | 20
Anaemia of malignant disease (Blood and lymphatic system disorders) | 42
Increased tendency to bruise (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Myelosuppression (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 4
Hypercalcaemia of malignancy (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 7
Hypophysitis (Endocrine disorders) | 1
Hypopituitarism (Endocrine disorders) | 1
Diplopia (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 4
Anal haemorrhage (Gastrointestinal disorders) | 1
Angular cheilitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 7
Enterocolitis (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 7
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 4
Disease progression (General disorders) | 2
Generalised oedema (General disorders) | 1
Influenza like illness (General disorders) | 2
Malaise (General disorders) | 5
Mucosal haemorrhage (General disorders) | 2
Mucosal inflammation (General disorders) | 4
Non-cardiac chest pain (General disorders) | 2
Oedema (General disorders) | 1
Pain (General disorders) | 4
Biliary obstruction (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 3
Contrast media allergy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Infusion related hypersensitivity reaction (Immune system disorders) | 3
Bacteraemia (Infections and infestations) | 1
Bacterial vaginosis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Candida infections (Infections and infestations) | 1
Biliary tract infection (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes oesophagitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pyuria (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Vulvovaginal candidiasis (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Amylase increased (Investigations) | 5
Bilirubin conjugated increased (Investigations) | 1
Blood albumin decreased (Investigations) | 4
Blood albumin increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatinine increased (Investigations) | 7
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
Blood urea increased (Investigations) | 2
Cell marker increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 5
Heart rate increased (Investigations) | 1
International normalised ratio increased (Investigations) | 2
Lipase increased (Investigations) | 6
Liver function test increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 6
Weight decreased (Investigations) | 7
Electrolyte imbalance (Metabolism and nutrition disorders) | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 4
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Sarcopenia (Musculoskeletal and connective tissue disorders) | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 8
Acute kidney injury (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Chromaturia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal injury (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Nipple pain (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Pruritus genital (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Milia (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin mass (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03833661/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT03833661/SAP_001.pdf